CLINICAL TRIAL: NCT06806917
Title: Twenty Years' Experience in Retroperitoneal Lymph Node Dissection for Testicular Cancer in a Tertiary Referral Center
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: RPLND-2021
Record Dates: First submitted 2025-01-10; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-12

CONDITIONS: Testicular Cancer
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to evaluate the oncologic and functional outcomes of RPLND as primary treatment (stage I and IIA-IIB with negative markers) or of residual masses after chemotherapy (PC-RPLND) in the treatment of patients with seminomatous and non-seminomatous.

In order to evaluate the role and the͛clinical impact of different surgical techniques of RPLND will be included patients treated with open, laparoscopic, and robot-assisted techniques

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the oncologic and functional outcomes of RPLND as primary treatment or residual masses after chemotherapy in the treatment of patients with seminomatous and nonseminomatous tumors.

In order to evaluate the role and clinical impact of different surgical techniques of RPLND will be included patients treated with open, laparoscopic, and robot-assisted techniques.

The study will be divided into two phases (a prospective and a retrospective phase):

* Phase 1 prospective is characterized by a multicenter prospective observational study international in which patients, competitively enrolled, undergo RPLND with open, laparoscopic or robot-assisted performed according to standard clinical practice from September 1, 2021 to October 31, 2026 and with 5-year follow-up.
* Retrospective Phase 2 is characterized by a multicenter retrospective international study involving the selection of patients who have already undergone RPLND, from January 2000 to December 2020 with a minimum follow-up of 12 months and data available from medical records, institutional databases, outpatient referrals or follow-up phone calls

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* RPLND of residual mass after chemotherapy in patient with testicular neoplasm seminomatous or nonseminomatous performed by open, laparoscopic, or robotic technique
* Primary RPLND for seminomatous or nonseminomatous testicular neoplasm of stage I or IIA-IIB with negative markers performed with open, laparoscopic or robotic technique
* RPLND performed by open, laparoscopic, or robotic technique for the treatment of tumors seminomatous or nonseminomatous chemiorefractory testicular tumors progressing after I and II line of chemotherapy
* Acquisition of informed consent

Exclusion criteria:

* Patient with comorbidities with contraindication to surgery
* Hemorrhagic diathesis

RETROSPECTIVE PHASE. Patients with the same inclusion and exclusion criteria as in the prospective phase and already undergoing RPLND surgery with open, laparoscopic, or robotic technique from January 2000 to December 2020 in the͛framework of the normal course of care with a minimum follow-up of 12 months. (estimated to include approximately 120 patients).

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Phase 1 prospective Patients selected for the prospective phase will undergo open, laparoscopic, or robotic according to the usual care pathway; follow-up visits will follow the normal clinic practice.
  Retrospective phase 2 Patients selected for the retrospective phase underwent open, laparoscopic, or robotic according to the normal course of care from January 2000 to December 2020 and have already been undergone follow-up postoperative examinations and examinations according to normal clinical practice with follow-up up of 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2031-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) and Recurrence-Free Survival (RFS) | through study completion, an average of 1 year
  To evaluate oncological outcomes, namely Overall Survival (OS) and Recurrence-Free Survival (RFS), of O-RPLND

SECONDARY OUTCOMES:
Intraoperative and postoperative complications | up to 3 months
  To describe intraoperative and postoperative complications, including ejaculatory disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Brunocilla, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- Italy (2):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - UO di Chirurgia Urologica della Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No